CLINICAL TRIAL: NCT05948046
Title: The Health-Related Quality of Life of the Patients With Symptomatic Convergence Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SGZX2203
Record Dates: First submitted 2023-06-21; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Myopia; Convergence Insufficiency
MeSH Terms: conditions — Myopia; Ocular Motility Disorders | interventions — Hospitals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training group: Patients with symptomatic convergence insufficiency who had received visual training
  Interventions: Behavioral: Visual training in hospital
- Not training group: Patients with symptomatic convergence insufficiency who had not received visual training

INTERVENTIONS:
Behavioral: Visual training in hospital — Completion of 1 session of standardized visual training
  Groups: Training group

SUMMARY:
This trial is an observational cohort study. Patients aged 8-15 years with symptomatic convergence insufficiency and 150 patients with symptomatic convergence insufficiency who had not received visual training were selected from the Tianjin Eye Hospital Optometry Center and received 1 course of visual training treatment. Self-assessment and other assessments were combined, and the patient and guardian questionnaires were collected. The EQ-5D-Y and CHU9D scales were used to evaluate Chinese patients' health-related quality of life with symptomatic convergence insufficiency. The feasibility of the EQ-5D-Y and CHU9D scales in assessing the health-related quality of life of Chinese patients with symptomatic convergence insufficiency was analyzed. To assess the effectiveness of visual training on visual symptoms and improvement of quality of life in patients with symptomatic convergence insufficiency

ELIGIBILITY:
Inclusion Criteria:

* 8~15 years old
* Monocular best corrected visual acuity at distance and near was more than 0.8
* Near exophoria 4Δ greater than distance exophoria
* NPC ≥ 6cm
* PFV ≤15△BO
* Stereogram ≤500 ''
* Score of CISS questionnaire ≥16 or COVD questionnaire≥20

Exclusion Criteria:

* present constant strabismus, nystagmus or vertical phoria at distance or near.
* developmental delay or ocular surgery
* Myopia≤ -6.00D, Hyperopia ≥ +5.00D, Astigmatism ≥ 4.00D
* Monocular Amplitude of accommodation<5D
* Other diseases except myopia

Ages: 8 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Adolescent patients with insufficient astringency
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in EuroQol five dimensions questionnaire(EQ-5D-5L) score | The changes between baseline and 3 months
  The EQ-5D-5L questionnaires were used to evaluate the quality of life scores of myopic patients.The health utility value can be calculated by the number of the answer to the question. 0 means death and 1 means complete health.
Changes in shortForm 6D(SF-6D) questionnaire score | The changes between baseline and 3 months
  The SF-6D questionnaires were used to evaluate the quality of life scores of myopic patients.The health utility value can be calculated by the number of the answer to the question. 0 means death and 1 means complete health.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No